CLINICAL TRIAL: NCT02027454
Title: A Study to Evaluate the Effect of GSK1265744 150mg Administered Orally Every 12h x 3 Doses on Cardiac Conduction as Assessed by 12-lead Electrocardiogram Compared to Placebo and a Single Oral Dose of Moxifloxacin
Brief Title: Study to Evaluate the Effect of GSK1265744 on Cardiac Conduction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 117009
Record Dates: First submitted 2013-11-07; First posted 2014-01-06 (Estimated); Last update posted 2014-06-16 (Estimated); Status verified 2014-06

CONDITIONS: Infection, Human Immunodeficiency Virus
Keywords: GSK1265744; HIV; placebo; cardiac repolarization; 12-lead ECG; moxifloxacin; QTc
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — cabotegravir; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Sequence 1 (Experimental): Participants in this arm will receive treatment A in period 1, treatment B in period 2 and treatment C in period 3. Where treatment A= Three doses of GSK1265744 150 mg (5 x 30mg tablets) every 12 hours. B= Three doses of GSK1265744 placebo (5 tablets) every 12 hours. C= A single dose of Moxifloxacin 400mg (one 400mg tablet).
  Interventions: Drug: GSK1265744; Drug: GSK1265744 matching placebo; Drug: Moxifloxacin
- Sequence 2 (Experimental): Participants in this arm will receive treatment A in period 1, treatment C in period 2 and treatment B in period 3. Where treatment A= Three doses of GSK1265744 150 mg (5 x 30mg tablets) every 12 hours. B= Three doses of GSK1265744 placebo (5 tablets) every 12 hours. C= A single dose of Moxifloxacin 400mg (one 400mg tablet).
  Interventions: Drug: GSK1265744; Drug: GSK1265744 matching placebo; Drug: Moxifloxacin
- Sequence 3 (Experimental): Participants in this arm will receive treatment B in period 1, treatment A in period 2 and treatment C in period 3. Where treatment A= Three doses of GSK1265744 150 mg (5 x 30mg tablets) every 12 hours. B= Three doses of GSK1265744 placebo (5 tablets) every 12 hours. C= A single dose of Moxifloxacin 400mg (one 400mg tablet).
  Interventions: Drug: GSK1265744; Drug: GSK1265744 matching placebo; Drug: Moxifloxacin
- Sequence 4 (Experimental): Participants in this arm will receive treatment B in period 1, treatment C in period 2 and treatment A in period 3. Where treatment A= Three doses of GSK1265744 150 mg (5 x 30mg tablets) every 12 hours. B= Three doses of GSK1265744 placebo (5 tablets) every 12 hours. C= A single dose of Moxifloxacin 400mg (one 400mg tablet).
  Interventions: Drug: GSK1265744; Drug: GSK1265744 matching placebo; Drug: Moxifloxacin
- Sequence 5 (Experimental): Participants in this arm will receive treatment C in period 1, treatment A in period 2 and treatment B in period 3. Where treatment A= Three doses of GSK1265744 150 mg (5 x 30mg tablets) every 12 hours. B= Three doses of GSK1265744 placebo (5 tablets) every 12 hours. C= A single dose of Moxifloxacin 400mg (one 400mg tablet).
  Interventions: Drug: GSK1265744; Drug: GSK1265744 matching placebo; Drug: Moxifloxacin
- Sequence 6 (Experimental): Participants in this arm will receive treatment C in period 1, treatment B in period 2 and treatment A in period 3. Where treatment A= Three doses of GSK1265744 150 mg (5 x 30mg tablets) every 12 hours. B= Three doses of GSK1265744 placebo (5 tablets) every 12 hours. C= A single dose of Moxifloxacin 400mg (one 400mg tablet).
  Interventions: Drug: GSK1265744; Drug: GSK1265744 matching placebo; Drug: Moxifloxacin

INTERVENTIONS:
Drug: GSK1265744 — White to slightly colored film coated tablet with unit dose strength of 30 mg and dose level of 150mg (5 tablets of 3 mg) administered orally every 12hours for 3 doses.
Drug: GSK1265744 matching placebo — GSK1265744 matching placebo tablets administered orally every 12hours for 3 doses (5 tablets per dose).
Drug: Moxifloxacin — Dull red, oblong, convex film coated tablets with unit dose strength of 400 mg administered orally as a single dose.

SUMMARY:
This study is being conducted to comply with the Food and Drug Administration (FDA) recommendation that all new non anti-arrhythmic drugs be assessed for cardiac repolarization effects through electrocardiographic evaluation. Therefore, this study will evaluate the effect of GSK1265744 on cardiac conduction as assessed by collection of twelve-lead continuous digital data in healthy adults. This study will evaluate the effect of three doses of GSK1265744 on the QT duration corrected for heart rate (QTc) interval as compared to placebo. Moxifloxacin will be used as a positive control in order to validate the sensitivity of the study in detecting QTc change. This study consists of three treatment periods (each separated by 21 day washout period) followed by follow-up visit 10 to 14 days post last dosing. The total duration of study including follow-up visit will be approximately 62 days. Approximately 42 subjects will be enrolled such that 34 subjects complete dosing and critical assessments.

ELIGIBILITY:
Inclusion Criteria:

* Male and females aged between 18 and 55 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* Body weight >=50 kilograms (kg) for men and >= 45 kg for women and body mass index (BMI) within the range 18.5-31.0 kg/meter^2 (inclusive).
* A female subject is eligible to participate if she is of: non-childbearing potential defined as pre-menopausal females with a documented tubal ligation, bilateral oophorectomy or hysterectomy [for this definition, "documented" refers to the outcome of the investigator's/designee's review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject's medical records]; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 milli international unit (MlU)/mililiter (m) and estradiol < 40 picogram/mL (<147 picomoles/L) is confirmatory] OR has only same-sex partners, when this is her preferred and usual lifestyle.
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods. This criterion must be followed from the time of the first dose of study medication until 21 days post-last dose.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria

* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 grams of alcohol: 12 ounces (360 mL) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GlaxoSmithKline (GSK) Medical Monitor, contraindicates their participation.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* Use of tobacco- or nicotine-containing products within 6 months prior to screening.
* A positive pre-study drug/alcohol screen.
* A positive test for human immuno virus antibody.
* Subjects with an alanine aminotransferase, alkaline phosphatase and bilirubin >=1.5xupper limit of normal (ULN) (isolated bilirubin <1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin >35%).
* The subject's systolic blood pressure is outside the range of 90 to140 milimeter of mercury (mmHg) or diastolic blood pressure is outside the range of 45 to 90mmHg or heart rate is outside the range of 50 to 100 beats per minute (bpm) for female subjects or 45 to 100 bpm for male subjects.
* Exclusion criteria for screening ECG (a single repeat is allowed for eligibility determination): are: male subjects with Heart rate <45 and >100 bpm and female subjects with heart rate <50 and >100 bpm, PR <120 and >220 milliseconds (msec), QRS duration <70 and >120 msec, QTcB >450 msec.

Evidence of previous myocardial infarction (Does not include ST segment changes associated with repolarization).

Any conduction abnormality (including but not specific to left or right complete bundle branch block, atrioventricular block [2nd degree or higher], Wolf Parkinson White syndrome).

Sinus Pauses > 3 seconds. Any significant arrhythmia which, in the opinion of the principal investigator and GSK medical monitor, will interfere with the safety for the individual subject.

Non-sustained or sustained ventricular tachycardia (>=3 consecutive ventricular ectopic beats).

* Where participation in the study would result in donation of blood or blood products in excess of 500mL within a 56 day period.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2014-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in QT duration corrected for heart rate by Fridericia's formulas (QTcF) for GSK1265744 | Baseline on Day -1 and Day 2 for Periods 1 - 3 (49 Days)
  QT interval is a measure of the time between the start of the Q wave and the end of the T wave in the heart's electrical cycle. QTcF interval will be obtained by digital electrocardiograms (ECG) obtained through 12 lead holter monitoring machine. Triplicate ECGs will be evaluated at each time point

SECONDARY OUTCOMES:
Change from baseline in QT duration corrected for heart rate by Bazett's formula (QTcB), individual corrected QTc ( QTci) values, QT, QRS, and PR for GSK1265744 | Baseline on Day -1 and Day 2 for Periods 1 - 3 (49 Days).
  Single ECG will be obtained at all timepoints during the study using an ECG machine that automatically measures PR (beginning of P wave to the beginning of the next QRS), QRS (beginning of Q to the end of the S wave), QT, and QTc intervals.
Change from baseline in heart rate (HR) for GSK1265744 | Baseline on Day -1 and Day 2 for Periods 1 - 3 (49 Days).
  Single ECGs will be obtained at all timepoints during the study using an ECG machine that automatically calculates the heart rate. Heart rate is defined as the number of heartbeats per unit of time, usually per minute.
Change from baseline in QTcF, QTcB, QTci, QT, QRS, and PR for placebo | Baseline on Day -1 and Day 2 for Periods 1 - 3 (49 Days).
  Single ECGs will be obtained at all timepoints during the study using an ECG machine that automatically calculates the QTcF, QTcB, QTCi, QT, QRS, PR intervals
Change from baseline in HR for placebo | Baseline on Day -1 and Day 2 for Periods 1 - 3 (49 Days).
  Single ECGs will be obtained at all timepoints during the study using an ECG machine that automatically calculates the heart rate. Heart rate is defined as the number of heartbeats per unit of time, usually per minute.
Change from baseline in QTcF, QTcB, QTci, QT, QRS, and PR for Moxifloxacin | Baseline on Day -1 and Day 2 for Periods 1 - 3 (49 Days).
  Single ECGs will be obtained at all timepoints during the study using an ECG machine that automatically calculates the QTcF, QTcB, QTCi, QT, QRS, PR intervals
Change from baseline in HR for Moxifloxacin. | Baseline on Day -1 and Day 2 for Periods 1 - 3 (49 Days).
  Single ECGs will be obtained at all timepoints during the study using an ECG machine that automatically calculates the heart rate. Heart rate is defined as the number of heartbeats per unit of time, usually per minute.
Composite of pharmacokinetic (PK) parameters for GSK1265744. | Blood samples will be collected at following time points: Day 1 pre-dose (15 minutes prior to first dose 1), and at Day 2 pre-dose (within 15 minutes prior to dosing), 0.5, 1, 2, 3, 4, 6.5, 8, 12, and 24 hours post last dose in each period.
  PK parameters include: area under the concentration-time curve from time zero to last time of quantifiable concentration (AUC[0-t]), area under the concentration-time curve from time zero extrapolated to infinite time (AUC[0-infinity]), maximum observed concentration (Cmax), time of occurrence of Cmax (tmax), apparent clearance following oral dosing (CL/F), apparent volume of distribution at steady state after oral administration (Vdz/F), and terminal phase half-life (t1/2) from plasma concentrations of GSK1265744.
Composite of PK parameters for Moxifloxacin (if needed). | Blood samples will be collected on Day 2 at pre-dose, 0.5, 1, 2, 3, 4, 6.5, 8, 12, and 24 hours post last dose in each period.
  PK parameters include: AUC (0-t), AUC (0-infinity), Cmax, tmax, CL/F, Vdz/f, and t1/2.
12-lead ECG as a measure of safety and tolerability. | Up to 62 days.
  12-lead ECGs will be performed with the subject in a semi-supine position having rested in this position for at least 10 minutes beforehand. ECGs will be obtained using an ECG machine that automatically calculates the QTcF, QTcB, QTCi, QT, QRS, PR intervals and HR.
Vital sign as a measure of safety and tolerability. | Up to 62 days.
  Vital sign measurement include: blood pressure and heart rate.
Number participants with adverse events as a measure of safety and tolerability. | Up to 62 days.
  AEs will be collected from the start of Study Treatment and until the follow-up contact.
Clinical laboratory parameters assessment as a measure of safety and tolerability. | Up to 62 days.
  Clinical laboratory assessment include: hematology, clinical chemistry, urinalysis and additional parameters as needed.
Change from baseline in QTcF, QTcB and QTci for GSK1265744 | Baseline on Day -1 and Day 2 for Periods 1 - 3 (49 Days).
  Single ECGs will be obtained at all timepoints during the study using an ECG machine that automatically calculates the QTcF, QTcB, and QTCi intervals.
Difference between GSK1265744 and placebo in terms of change from baseline in QTcF, QTcB and QTci. | Baseline on Day -1 and Day 2 for Periods 1 - 3 (49 Days).
  Difference between GSK12657744 and placebo in terms of change from baseline in QTcF, QTcB and QTci will be measured to characterize pharmacodynamic (PD) relationship between exposure of GSK1265744 and changes in QTcF, QTcB and QTci
Plasma concentration profile as assessed from composite of PK parameters of GSK1265744. | Blood samples will be collected at following time points: Day 1 pre-dose (15 minutes prior to first dose 1), and at Day 2 pre-dose (within 15 minutes prior to dosing), 0.5, 1, 2, 3, 4, 6.5, 8, 12, and 24 hours post last dose in each period.
  Plasma concentration profile of GSK1265744 will be assessed to characterize PK/PD relationship between exposure of GSK1265744 and changes in QTcF, QTcB and QTci. PK parameters to be assessed for plasma concentration profile are: area under the concentration-time curve from zero to 24 hours (AUC [0-24]), AUC (0-t), AUC (0-infinity), and Cmax.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Overland Park, Kansas, United States